CLINICAL TRIAL: NCT03430986
Title: A Randomized, Multicenter, "No-Treatment" Control Study to Evaluate the Safety and Effectiveness of JUVÉDERM® VOLUMA® With Lidocaine Injectable Gel for the Improvement of Volume and Aesthetic Appearance of the Nose in Chinese Adults
Brief Title: Safety and Effectiveness of JUVÉDERM® VOLUMA® With Lidocaine for Improvement of Volume and Aesthetic Appearance of the Nose in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1894-701-008
Record Dates: First submitted 2018-02-02; First posted 2018-02-13 (Actual); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Nose Enhancement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JUVÉDERM® VOLUMA® with Lidocaine (Experimental): Participants were treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel during the 24-week Control Period. Participants were eligible for touch-up treatment 8 weeks after the initial treatment, if applicable. Follow-up continued in the 24-week Post-Control period.
  Interventions: Device: JUVÉDERM® VOLUMA® with Lidocaine
- No-treatment Control (Experimental): Participants received no treatment during the 24-week Control Period. After 24 weeks, participants had the option of treatment with JUVÉDERM® VOLUMA® with Lidocaine Injectable Gel in the nose area during the 24-week Post-Control period and were eligible for touch-up treatment 8 weeks after the initial treatment, if applicable.
  Interventions: Device: JUVÉDERM® VOLUMA® with Lidocaine; Other: No-treatment control

INTERVENTIONS:
Device: JUVÉDERM® VOLUMA® with Lidocaine — Treatment with JUVÉDERM® VOLUMA® with Lidocaine injectable gel with optional treatment 8 weeks later.
Other: No-treatment control — No treatment during the control period.
  Arms: No-treatment Control

SUMMARY:
The purpose of this study is to determine whether VOLUMA with Lidocaine is safe and effective for the improvement of volume and aesthetic appearance of the nose in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Is not satisfied with his/her aesthetic appearance due to structural features of his/her nose and assessed as either "dissatisfied" or "very dissatisfied" by using the 5-point Nose Satisfaction Scale (NSS)
* Requires a total volume of at least 0.5 mL but not exceeding 3.0 mL of VOLUMA with Lidocaine for initial and touch-up treatment combined, and treatment to the nasal dorsum is mandatory to achieve an aesthetic improvement in the subject's nose appearance, in the Treating Investigator (TI's) opinion
* Has a reasonable treatment goal for aesthetic improvement in nose, in the TI's opinion. Participant and TI have aligned the treatment goals.

Exclusion Criteria:

* Has a small, shallow nose such that the volume of filler implant needed to create the desired dorsal height is in excess of the ability of the skin and soft tissue to expand and accommodate the implant
* Has active autoimmune disease
* Is on a concurrent regimen of lidocaine or structurally-related local anesthetics (eg, bupivacaine)
* Is on an ongoing regimen of anti-coagulation therapy (eg, warfarin)
* Within 10 days of undergoing study device injection, is on an ongoing regimen of medications (eg, aspirin or ibuprofen) or other substances (eg, high doses of Vitamin C or Vitamin E or herbal supplements with garlic, gingko biloba, or ginseng) known to increase coagulation time, or is currently menstruating (study treatment may be delayed as necessary to accommodate menstrual period cessation and/or anticoagulation washout interval)
* Has participated in any clinical trials within 4 weeks prior to signing the informed consent form (ICF) or is planning to participate in another clinical trial during the course of this study
* Females who are pregnant, nursing, or planning a pregnancy during the course of the study. Females of childbearing potential who have a positive pregnancy test result during screening. Females who intend to breastfeed during the study. Females of childbearing potential who are unwilling to use birth control measures during the full course of the study. Birth control measures include oral contraceptives (stable) use for 2 or more cycles prior to screening), intrauterine devices, hormonal injections, hormonal implants, bilateral tube ligation, vasectomy, condom or diaphragm plus either contraceptive sponge, foam, or jelly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Zhang, Study Director — Allergan
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Beijing, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Beijing, Wuhan

RESULTS

PARTICIPANT FLOW:
Period: 24-week Control Period
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine
Started | 42 | 122
Treated as Randomized | 42 | 120
Completed | 34 | 118
Not Completed | 8 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Participant | 5 | 0
Not completed — Protocol Deviation | 0 | 2
Period: 24-week Post-Control Period
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine
Started | 31 (Not all participants received the Optional Treatment.) | 118
Completed | 30 | 116
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Participant | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) included all participants who were randomized to study treatment and received at least one study device treatment and completed at least 1 effectiveness assessment (treatment group) and participants who were randomized to no treatment and complete at least 1 effectiveness assessment (control group).
Groups:
- Total: Total of all reporting groups
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine | Total
Number analyzed (Participants) | 37 | 120 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.95) | 32.0 (10.42) | 31.3 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 112 | 147
  Male | 2 | 8 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 37 | 120 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 37 | 120 | 157
Region of Enrollment [Count of Participants; unit: Participants]
  China | 37 | 120 | 157

OUTCOME MEASURES:

1. Primary Outcome: Volume Change From Baseline in the Nose Area
Description: Volume of the nose was calculated by digital analysis of each participant's 3-dimensional (3D) images. A mixed-effects model for repeated measures (MMRM) was used for analysis. A positive change from Baseline indicates improvement. An analysis model was created by Canfield Scientific, only volume changes are available. Actual Baseline values are not available.
Time Frame: Baseline (Last value prior to treatment for the treatment group and last value prior to randomization for control group) to Week 24
Population: mITT Population included all participants who are randomized to study treatment and received at least one study device treatment and completed at least 1 effectiveness assessment (treatment group) and participants who are randomized to no treatment and complete at least 1 effectiveness assessment (control group).
Measure: Least Squares Mean (Standard Error); unit: cubic centimeters (cc)
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine
Number analyzed (Participants) | 37 | 120
cubic centimeters (cc) | -0.005 (0.1381) | 2.032 (0.0764)
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLUMA® With Lidocaine; Test type: Superiority; p < 0.0001, MMRM; MMRM included treatment, timepoint, treatment-by-timepoint interaction as fixed effect using an unstructured covariance matrix; Least Squares (LS) Mean Difference = 2.037, 95% CI 2-sided [1.726 to 2.349], Standard Error of Mean 0.1578

2. Secondary Outcome: Percentage of Participants Where the Evaluating Investigator Noted "Improved" or "Much Improved Using the Global Aesthetic Improvement Scale (GAIS)
Description: The Evaluating Investigator assessed the aesthetic improvement of the nose using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who the Evaluating Investigator assessed as 2=much improved or 1=improved is reported.
Time Frame: Week 24
Population: mITT Population included all participants who are randomized to study treatment and received at least one study device treatment and completed at least 1 effectiveness assessment (treatment group) and participants who are randomized to no treatment and complete at least 1 effectiveness assessment (control group). Participants analyzed are the number of participants with available data at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine
Number analyzed (Participants) | 32 | 117
percentage of participants | 18.8 [7.2 to 36.4] | 87.2 [79.7 to 92.6]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLUMA® With Lidocaine; Test type: Superiority; p < 0.0001, Fisher Exact; 2-sided test comparing responder rate between treatment group and control group; Percentage difference = 68.4, 95% CI 2-sided [50.0 to 82.4]

3. Secondary Outcome: Percentage of Participants Who Noted "Improved" or "Much Improved" as Assessed by the Participant Using the GAIS in the Treatment Group
Description: The participant assessed the aesthetic improvement of the nose using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who assess themselves as 2=much improved or 1=improved is reported.
Time Frame: Week 24
Population: mITT Population included all participants who are randomized to study treatment and received at least one study device treatment and completed at least 1 effectiveness assessment (treatment group). Participants analyzed is the number of participants with available data at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JUVÉDERM® VOLUMA® With Lidocaine
Number analyzed (Participants) | 117
percentage of participants | 91.5 [84.8 to 95.8]

4. Secondary Outcome: Percentage of Participants Who Noted "Satisfied" or "Very Satisfied" With Treatment Outcome on the Nose Satisfaction Scale (NSS) in the Treatment Group
Description: The participant used the 5-point NSS to assess the treatment outcome of the nose where: +2=very satisfied, +1=satisfied, 0=neutral (neither satisfied or dissatisfied), -1=dissatisfied and -2= very dissatisfied. The percentage of participants who assessed themselves as +2=Very Satisfied or +1=Satisfied is reported.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JUVÉDERM® VOLUMA® With Lidocaine
Number analyzed (Participants) | 117
percentage of participants | 95.7 [90.3 to 98.6]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) in the Control Period
Description: An AE is any untoward medical occurrence in a patient or a participant using an investigational drug, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: 24 Weeks
Population: Safety Population included all randomized participants who received VOLUMA treatment in the Control Period (CP) or who did not receive VOLUMA treatment in the CP and had at least 1 follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | No-treatment Control | JUVÉDERM® VOLUMA® With Lidocaine
Number analyzed (Participants) | 37 | 120
Participants | 17 | 43

ADVERSE EVENTS:
Time Frame: JUVÉDERM® VOLUMA® with Lidocaine Treatment group: 48 Weeks after last treatment (Up to 56 Weeks); No-treatment Control group: no treatment for 24 weeks then 24 weeks following last treatment (Up to 32 Weeks)
Description: Number of participants for All-cause Mortality included all randomized participants. Number of participants for Serious Adverse Events and Adverse Events is based on the Safety Population that included all randomized participants who received VOLUMA treatment in the CP or who did not receive VOLUMA treatment in the CP and had at least 1 follow-up assessment or participants in the VOLUMA Optionally Treated arm who received treatment.
Groups:
- No-treatment Control (Control Period): Participants who received no treatment during the 24-week Control Period.
- JUVÉDERM® VOLUMA® With Lidocaine (Control Period): Participants were treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel to the nose area during the 24-week Control Period. Participants were eligible for touch-up treatment 8 weeks after the initial treatment, if applicable.
- VOLUMA Initially Treated (Post-Control Period): Participants in the 24-week Post-Control Period who were treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel during the 24-week Control Period.
- VOLUMA Optionally Treated (Post-Control Period): Participants in the 24-week Post-Control Period who received no treatment in the 24-week Control Period then were treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel with an optional treatment 8 weeks later, if applicable
Arm/Group | No-treatment Control (Control Period) | JUVÉDERM® VOLUMA® With Lidocaine (Control Period) | VOLUMA Initially Treated (Post-Control Period) | VOLUMA Optionally Treated (Post-Control Period)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/122 | 0/118 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/120 | 2/118 | 1/31
Other Adverse Events (participants affected / at risk) | 12/37 | 20/120 | 23/118 | 10/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (Control Period) (N=37) | JUVÉDERM® VOLUMA® With Lidocaine (Control Period) (N=120) | VOLUMA Initially Treated (Post-Control Period) (N=118) | VOLUMA Optionally Treated (Post-Control Period) (N=31)
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (Control Period) (N=37) | JUVÉDERM® VOLUMA® With Lidocaine (Control Period) (N=120) | VOLUMA Initially Treated (Post-Control Period) (N=118) | VOLUMA Optionally Treated (Post-Control Period) (N=31)
Nasopharyngitis (Infections and infestations) | 5 | 10 | 12 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 8 | 10 | 3
Periodontitis (Infections and infestations) | 2 | 0 | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2
Pyrexia (General disorders) | 1 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT03430986/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03430986/SAP_001.pdf